CLINICAL TRIAL: NCT07040267
Title: Investigation of the Effect of Smartphone Addiction on the Biomechanical Properties of Thumb Muscles and Thumb Sensory Sensitivity in University Students
Brief Title: Smartphone Addiction on the Biomechanical Properties of Thumb Muscles and Thumb Sensory Sensitivity
Status: Recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, ESRA PEHLIVAN, Principal Investigator, Saglik Bilimleri Universitesi
Other Study IDs: Smartphone Addiction& Thumb-1
Record Dates: First submitted 2025-06-18; First posted 2025-06-27 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Smartphone Addiction; Thumb Injury
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Smartphone-Addicted Group: This group will consist of university students who will be identified as addicted to smartphones based on their scores on the Smartphone Addiction Scale - Short Version (SAS-SV). Participants scoring above the cut-off threshold will be assigned to this group. Weekly screen time will also be recorded.
  Interventions: Diagnostic Test: Thumb evaluations
- Non-Addicted Control Group: This group will consist of university students who will be identified as not addicted to smartphones based on their SAS-SV scores, scoring below the determined cut-off point. Weekly screen time will also be recorded.
  Interventions: Diagnostic Test: Thumb evaluations

INTERVENTIONS:
Diagnostic Test: Thumb evaluations — There is no therapeutic or experimental intervention in this study. All procedures will be limited to diagnostic evaluations. The study will include non-invasive biomechanical and sensory assessments to compare the thumb muscle characteristics and sensory discrimination between smartphone-addicted and non-addicted university students.
  Specifically, muscle tone, stiffness, and elasticity will be measured using the MyotonPro™ device, and thumb sensory sensitivity will be evaluated using a Baseline Aesthesiometer with a two-point discrimination test. These assessments will be conducted during a single laboratory visit and will not involve any treatment, medication, or behavioral intervention.
  This is a purely observational study aimed at identifying potential associations between smartphone usage patterns and thumb neuromuscular or sensory changes.

SUMMARY:
This study will aim to assess the effects of smartphone addiction on thumb muscle biomechanics and sensory sensitivity among university students. The research will investigate whether excessive smartphone use leads to significant differences in muscle tone, stiffness, elasticity, and sensory discrimination capabilities.

DETAILED DESCRIPTION:
This will be a prospective, non-randomized, controlled observational study designed to examine the impact of smartphone addiction on the neuromuscular and sensory function of the thumbs. A total of 36 university students aged 18 to 30 will be recruited and categorized into two groups based on their scores from the Smartphone Addiction Scale - Short Version (SAS-SV): addicted and non-addicted.

Participants' weekly screen times will be recorded, and the smartphone applications used will be categorized. The MyotonPro™ device will be used to measure the biomechanical properties of three thumb muscles (abductor pollicis brevis, flexor pollicis brevis, and opponens pollicis) in both hands. Sensory function will be assessed bilaterally using the Baseline Aesthesiometer via two-point discrimination testing.

This study will evaluate whether significant biomechanical or sensory changes are observable among addicted users compared to non-addicted users, and whether screen time is correlated with any muscular or sensory outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-30 years
* Currently enrolled university students
* Regular smartphone users

Exclusion Criteria:

* Presence of systemic, chronic, or neuromuscular disorders
* History of upper limb surgery or trauma
* Neurological or orthopedic conditions affecting upper extremities
* Subcutaneous fat over target muscles >20 mm
* Presence of wounds or burns on the measurement area

Ages: 18 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: The study population will consist of university students aged 18 to 30 years who are regular smartphone users. Participants will be recruited from a university setting and will voluntarily participate in the study after providing written informed consent. Both male and female students will be eligible.
  Participants will be assigned to one of two groups-smartphone-addicted or non-addicted-based on their scores on the Smartphone Addiction Scale - Short Version (SAS-SV). Only healthy individuals without any systemic, neurological, musculoskeletal, or upper extremity disorders will be included. The study will focus on a relatively homogeneous group of young adults to examine the early neuromuscular and sensory impacts of smartphone usage.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
MyotonPro™ Muscle Assessment | Baseline
  This device will be used to assess muscle tone, stiffness, and elasticity in the abductor pollicis brevis, opponens pollicis, and flexor pollicis brevis muscles of both hands. Measurements will be performed with the participant in a standardized seated position.

SECONDARY OUTCOMES:
Baseline Aesthesiometer Sensory Assessment | Baseline
  This instrument will be used to evaluate thumb sensory sensitivity through two-point discrimination testing on both hands. Participants will be blindfolded during the procedure and tested at the distal phalanx of the thumb.
Smartphone Addiction Scale - Short Version (SAS-SV) | Baseline
  The Smartphone Addiction Scale - Short Version (SAS-SV) is a validated self-report questionnaire developed to assess the risk of smartphone addiction, particularly in adolescents and young adults. It consists of 10 items, each rated on a 6-point Likert scale ranging from 1 (strongly disagree) to 6 (strongly agree). The total score ranges from 10 to 60, with higher scores indicating a greater risk of smartphone addiction.

CONTACTS AND LOCATIONS:
Locations (1):
- Esra Pehlivan, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided